CLINICAL TRIAL: NCT00611507
Title: A Phase II Study of Oxaliplatin in Association With 5FU and Folinic Acid in the Treatment of Subjects With Non-Surgical or Advanced Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Juan Carlos Gomez/Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8107
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin, 5-Fluorouracil — 5FU 500 mg/m² per week in IV bolus infusion during 30 min AF 20mg/m²/week in infusion, during 10-20 minutes prior 5FU infusion; Eloxatin 85 mg/m² as IV infusion 2-6 hours, every 2 weeks. Three weeks of treatment, one week rest.
  Other Names: Eloxatin, 5FU

SUMMARY:
This phase II trial will evaluate, in first line advanced or metastatic gastric cancer, the efficacy and tolerance of another oxaliplatin, 5FU bolus combination already tested in advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric or gastroesophagic junction adenocarcinoma
* Measurable disease at least in a unidimensional manner. If a unique metastasis constitutes the only disease symptom, histological confirmation will be required
* Metastatic or locally non-surgical primary gastric cancer
* Recurrent gastric cancer after local and/or systemic treatment with a post-surgical period of at least 4 weeks, a post-adjuvant chemotherapy period or a neo-adjuvant chemo-radiotherapy of at least 6 months
* Serum bilirubin< 2 mg/dl
* Serum creatinine < or =to 2 times normal superior limit
* Absolute neutrophil count > or =to 2000/dl
* Platelet count > or =to 100000/dl
* Hemoglobin > or =to 10 g/dl
* AST/ALT < or =to 2.5 times normal superior institutional limit
* Alkaline phosphatase < or =to 5 times the normal superior institutional limit
* Age > 18 years
* Performance Status ECOG 0-2
* Written informed consent signed and dated

Exclusion Criteria:

* Symptomatic sensory peripheral neuropathy
* Uncontrolled concomitant disease.(e.g. severe diabetes mellitus, arterial hypertension)
* Any other malignancy diagnosed within 5 years previous to the gastric cancer, with the exception of " in situ " cervix carcinoma or non-melanoma skin cancer
* Concomitant anti-tumoral treatment
* Cerebral metastases
* Unstable heart disease, even though under treatment
* Myocardial infarction within the last 6 months
* Pregnancy or nursing (or women in reproductive life without adequate contraception)
* Significant neurological or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Response rate - RECIST criteria (unidimensional) | During the study conduct

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Gomez, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bogotá, Colombia